CLINICAL TRIAL: NCT01052584
Title: Ethiopia In-vivo Efficacy Study 2009: Evaluating the Efficacy of Artemether-lumefantrine for the Treatment of Uncomplicated Plasmodium Falciparum Infection and Either Artemether-lumefantrine or Chloroquine for P. Vivax Infection
Brief Title: Ethiopia Malaria Therapeutic Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Columbia University (Other)
Responsible Party: Jimee Hwang/ Medical Epidemiologist, CDC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCZVED-5628
Record Dates: First submitted 2010-01-17; First posted 2010-01-20 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Malaria
Keywords: malaria; therapeutic efficacy; in vivo; artemether lumefantrine; coartem; chloroquine; Plasmodium falciparum; Plasmodium vivax
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chloroquine-P. vivax (Experimental): P. vivax randomized to receive chloroquine 3-day regimen
  Interventions: Drug: Chloroquine- P. vivax
- Artemether-Lumefantrine: P. vivax (Experimental)
  Interventions: Drug: Artemether-Lumefantrine: P. vivax
- Artemether-lumefantrine: P. falciparum (Experimental): administered twice daily for three days as tablets containing 20 mg of artemether plus 120 mg of lumefantrine in a fixed dose combination at a dosage
  Interventions: Drug: Artemether-lumefantrine: P. falciparum

INTERVENTIONS:
Drug: Chloroquine- P. vivax — Total of 25mg base per kg over 3 days (10 mg base/kg on Days 1 and 2, and 5 mg base/kg on Day 3)
  Arms: Chloroquine-P. vivax
Drug: Artemether-Lumefantrine: P. vivax — administered twice daily for three days as tablets containing 20 mg of artemether plus 120 mg of lumefantrine in a fixed dose combination at a dosage
  Arms: Artemether-Lumefantrine: P. vivax
Drug: Artemether-lumefantrine: P. falciparum — administered twice daily for three days as tablets containing 20 mg of artemether plus 120 mg of lumefantrine in a fixed dose combination at a dosage
  Arms: Artemether-lumefantrine: P. falciparum

SUMMARY:
In this stdy, patients aged above 6 months with symptomatic malaria presenting to health centers will be enrolled for treatment with artemether-lumefantrine for P. falciparum infection, and either artemether-lumefantrine or chloroquine for P. vivax infection. Clinical, parasitologic, and hematologic parameters will be monitored for P. falciparum and P. vivax infection over a 42-day follow-up period, which will be used to evaluate drug efficacy. Results from this research study will be used to assist Ethiopia in assessing their current national malaria drug policies.

DETAILED DESCRIPTION:
Following the rapid development of significant drug resistance of Plasmodium falciparum (Pf) to chloroquine and then sulfadoxine-pyrimethamine (the first line therapy in Ethiopia 1998-2004), artemether- lumefantrine (Coartem or AL) was adopted as first line therapy in Ethiopia in 2004. According to the current national malaria diagnosis and treatment guidelines, first-line treatment for uncomplicated falciparum infection is AL. First-line treatment for Plasmodium vivax (Pv) is with chloroquine (CQ) alone without primaquine therapy in malarious areas. For all clinical infection without laboratory confirmation, AL which is effective against both Pf and Pv is the first-line treatment. Thus, in Ethiopia, where treatment for malaria without laboratory confirmation occurs frequently, Pv is often treated with AL as the standard of care. Furthermore, World Health Organization (WHO) recommends AL for the treatment of Pv, where AL has been adopted as first-line treatment for Pf. Now with wide-spread use of AL and CQ, we propose to conduct an antimalarial efficacy study to monitor the effectiveness of these therapies in Ethiopia and to determine how efficacious these drugs remain. This information will inform future policy changes with respect to appropriate antimalarial strategies.

The simplest and most universally accepted measure of testing for antimalarial drug treatment efficacy, the standardized procedures outlined in the World Health Organization Assessment and monitoring of antimalarial drug efficacy for the treatment of uncomplicated falciparum malaria and the WHO Monitoring antimalarial drug resistance, will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Slide-confirmed infection with P. falciparum, with parasitemia of 1,000-100,000 asexual forms/ μl or slide confirmed infection with P. vivax with > 250 asexual forms/ μl
* Lives within 20 km of the enrolling health facility
* Weight ≥ 5.0 kg
* Axillary temperature ≥ 37.5º C or history of fever during the previous 24 or 48 hours for P. falciparum and P. vivax infection, respectively
* Patient or caregiver agrees to all blood draws and return visits.

Exclusion Criteria:

* General danger signs or symptoms of severe malaria
* Signs or symptoms of severe malnutrition, defined as weight-for-age ≤ 3 standard deviations below the mean (NCHS/WHO normalized reference values;
* Slide confirmed infection with any other Plasmodium spp. besides falciparum/vivax or mixed plasmodium infection
* Severe anemia, defined as Hg < 5 g/dl
* Known hypersensitivity to any of the drugs being evaluated
* Presence of febrile conditions caused by diseases other than malaria
* Serious or chronic medical condition (cardiac, renal, hepatic diseases, sickle cell disease, HIV/AIDS)
* Pregnant or breastfeeding women.
* Children weighing less than 5 kilograms.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Determine Early Treatment Failures, Late Clinical Failures, Late Parasitological Failures, or Adequate Clinical and Parasitological Response during 28 days of follow-up for P. falciparum. Measure the treatment failure of AL and CQ for P. vivax | 28 days

SECONDARY OUTCOMES:
Determine Early Treatment Failures, Late Clinical Failures, Late Parasitological Failures, or Adequate Clinical and Parasitological Response during 42 days of follow-up for P. falciparum. Measure the treatment failure of AL and CQ for P. vivax durin | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Jimee Hwang, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- Ethiopia (2):
  - DebreZeit Malaria Center, Debrezeit, Oromiya
  - Bulbula Health Center, Zeway, Oromiya

REFERENCES:
- [Derived] Hwang J, Alemayehu BH, Reithinger R, Tekleyohannes SG, Takele Teshi, Birhanu SG, Demeke L, Hoos D, Melaku Z, Kassa M, Jima D, Malone JL, Nettey H, Green M, Poe A, Akinyi S, Udhayakumar V, Kachur SP, Filler S. In vivo efficacy of artemether-lumefantrine and chloroquine against Plasmodium vivax: a randomized open label trial in central Ethiopia. PLoS One. 2013 May 22;8(5):e63433. doi: 10.1371/journal.pone.0063433. Print 2013. PMID 23717423
- [Derived] Hwang J, Alemayehu BH, Hoos D, Melaku Z, Tekleyohannes SG, Teshi T, Birhanu SG, Demeke L, Gobena K, Kassa M, Jima D, Reithinger R, Nettey H, Green M, Malone JL, Kachur SP, Filler S. In vivo efficacy of artemether-lumefantrine against uncomplicated Plasmodium falciparum malaria in Central Ethiopia. Malar J. 2011 Jul 28;10:209. doi: 10.1186/1475-2875-10-209. PMID 21798054